CLINICAL TRIAL: NCT05520086
Title: Phase IIa Multicenter Clinical Trial to Determine the Feasibility and Safety of the Use of Adipose-derived Mesenchymal Stem Cells (ASC) in the Treatment of Patients With Cicatricial Conjunctivitis Associated With Lyell's Syndrome, Stevens-Johnson Syndrome and Pemphigoid of the Mucous Membranes With Ocular Involvement.
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of Cell Therapy in Patients With Cicatricial Conjuntivitis.
Acronym: CELOPHIN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CELOPHIN
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Conjunctivitis; Stevens-Johnson Syndrome; Lyell Syndrome; Pemphigoid
MeSH Terms: conditions — Stevens-Johnson Syndrome; Pemphigoid, Bullous

STUDY DESIGN:
Intervention Model Description: 2 consecutive cohorts will be included in order of recruitment. the first 10 patients will receive 1 single dose and the second 10 patients will receive 2 doses separated by 15 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose Allogenic Adiposse derived mesenchimal stem cells (Experimental): Allogenic Adiposse derived mesenchimal stem cells (MSC) Dose: 12,5 million cells
  Interventions: Drug: Single Dose
- Double dose Allogenic Adiposse derived mesenchimal stem cells (Experimental): Allogenic Adiposse derived mesenchimal stem cells (MSC) Dose: 12,5 million cells at day 0 and 12,5 million cells at day 14
  Interventions: Drug: Double Dose

INTERVENTIONS:
Drug: Single Dose — Single Dose: Administration of 12,5 million allogeneic mesenchymal stem cells derived from adipose tissue by subcnjunctival injection and topical conjunctival injection.
  Arms: Single dose Allogenic Adiposse derived mesenchimal stem cells
Drug: Double Dose — Repetead Dose: Administration of 2 doses, separated by 14 days, of 12,5 million allogeneic mesenchymal stem cells derived from adipose tissue by subcnjunctival injection and topical conjunctival injection.
  Arms: Double dose Allogenic Adiposse derived mesenchimal stem cells

SUMMARY:
A phase IIa, open label, non controlled clinical trial to assess the feasibility and safety of allogeneic adipose-derived mesenchymal stem cells (ASC) in the treatment of cicatricial conjunctivitis associated with Lyell's syndrome, Stevens-Johnson's syndrome and mucous membrane pemphigoid with ocular involvement

DETAILED DESCRIPTION:
A multicentre, nationwide clinical trial will be performed. 20 patients fulfilling eligibility criteria will be included in two different dose level cohorts: the first 10 patients included will receive a single cell application and the remainder 10 will be administered 2 cell applications separated by 15 days.

The investigational drug consists of locally administered, expanded, allogeneic adipose-derived adult mesenchymal stem cells (ASCs), at a dose of 5 million cells per ml (0,5 ml to be infused per quadrant)

Study cronogram: recruitment is estimated to take 8 months, and follow-up period will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Diagnosis of ocular pemphigoid in Foster stages I-IIcIIIb (2) or diagnosis of recurrent chronic or episodic inflammation accompanied by cicatricial conjunctivitis of the mucous membranes with ocular involvement after the acute phase of Stevens-Johnson Syndrome or Lyell Syndrome with insufficient disease control or inaceptable toxicity or impossibility to administer usual care treatments (according to physician or patient criteria)
3. In the case of women of childbearing age, who are willing to use an effective contraceptive method during the period of participation in the study
4. Consent to participate and signature of the informed consent

Exclusion Criteria:

1. Signs of active infection on the ocular surface.
2. History of neoplasms in the last 5 years. except for epithelial basal or squamous cell carcinoma
3. Allergy to local anesthetics
4. Patients who have participated in another clinical trial with medication during the 90 days prior to signing the IC
5. Medical or psychiatric illness of any kind that, in the opinion of the investigator, may be a reason for exclusion from the study.
6. Congenital or acquired immunodeficiencies.
7. Major surgery or serious trauma of the subject in the semester prior to signing the IC.
8. Pregnant or lactating women.
9. Impossibility or refusal to carry out the follow-up required in the study by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-11-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of complications | Through study completion, an average of 3 years
  Percentage of complications related to anesthesia, administration of investigational medicinal product and postoperative period.

SECONDARY OUTCOMES:
Signs improvement | At 7 days (and 21 days in the 2-dose group), 4 weeks, 12 weeks, 24 weeks and 52 weeks
  Changes from baseline in scarring conjunctivitis rating scale
Symptom improvement | At 7 days (and 21 days in the 2-dose group), 4 weeks, 12 weeks, 24 weeks and 52 weeks
  Changes from baseline in Ocular Surface Disease Index (OSDI) questionnaire (0-48). The lower the rate obtained in the score, better the outcome.
Visual acuity improvement | At 7 days (and 21 days in the 2-dose group), 4 weeks, 12 weeks, 24 weeks and 52 weeks
  Changes from baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) (0-1,2).
  The higher the rate obtained in the score, better the outcome.
changes in quality of life | At 7 days (and 21 days in the 2-dose group), 4 weeks, 12 weeks, 24 weeks and 52 weeks
  Changes from baseline using the specific National Eye Institute-Visual Function Questionnaire 25 (NEI-VFQ-25) (0-100). The value of 0 is the lowest and 100 the best possible
evolution of the conjunctival flora | At 7 days (and 21 days in the 2-dose group), 4 weeks, 12 weeks, 24 weeks and 52 weeks
  variation in the number and type of microorganisms in the conjunctival exudates, performing cultures and PCR herpes viridae

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Alejandre Alba, Principal Investigator — Hospital Fundación Jiménez Diaz
Locations (8):
- Spain (8):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital General La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Instituto Oftalmológico Fernández - Vega, Oviedo, Principality of Asturias
  - Hospital La Arruzafa, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundación Jiménez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No